CLINICAL TRIAL: NCT06882213
Title: Unlocking Trunk Potential After Stroke: A Novel Approach Combining Transcranial Direct Current Stimulation and Core Stability Exercise
Brief Title: Combining Transcranial Direct Current Stimulation and Core Stability Exercise on Trunk in Stroke Patient
Acronym: TCDC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Lecturer of Physical therapy, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Transcranial Direct Current
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): will receive simultaneously a combination of transcranial direct current stimulation combined with core stability exercise.
  Interventions: Other: transcranial direct current stimulation; Other: core stability exercise.
- Control group (Active Comparator): will receive core stability exercise.
  Interventions: Other: core stability exercise.

INTERVENTIONS:
Other: transcranial direct current stimulation — transcranial direct current stimulation
  Arms: Study Group
Other: core stability exercise. — core stability exercise.

SUMMARY:
To evaluate the effects of the combining transcranial direct current stimulation with core stability exercises on trunk performance in poststroke hemiparetic patients, the secondary outcome is to evaluate the balance and the functional performance of the participants.

DETAILED DESCRIPTION:
This study will conduct to 60 male and female patients with post stroke hemiparesis with age ranged between 55 to 70 years, the patients will be categorized to two equal groups.

* Group A (study group): will receive simultaneously a combination of transcranial direct current stimulation combined with core stability exercise.
* Group B (control group): will receive core stability exercise. All patients will be assessed for trunk performance, balance, and functional performance before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are ≥ 55 years old of both sex, had a first-time right or left stroke within the preceding six months that damaged the cerebral cortex verified by (computed tomography or MRI report, neurological examination, and medical chart).
* Patients can stand and walk independently.
* Modified Ashworth Scale (MAS) of upper limb muscle ≤ 1+.
* All the patients received a conventional physiotherapy program in the acute stage and post-discharge from the hospital.
* None of the patients participated in any other study or placebo

Exclusion Criteria:

* Patients with neurological or orthopedic problems, paralysis neglect, behavioral abnormalities, dementia any shoulder dysfunction before or post-stroke (dislocation or subluxation), or those who using upper limb splints.
* Recurrent strokes or hemiparesis due to other neurological causes rather than stroke eg .(Brain tumor).
* Obesity (BMI ≥ 30 kg/m2).

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale (TIS). | up to 8 weeks
  trunk performance will be assessed by Trunk Impairment Scale (TIS).
Berg Balance Scale | up to 8 weeks
  Balance will be assessed by berg balance scale, the balance score ranges from 0 to 56, with lower scores indicating increased risk of balance loss and higher scores indicating improved functional mobility. Time up and go test (TUG)n Score < 10 seconds = normal < 20 seconds = good mobility; can walk outside alone; does not require a walking aid < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid

CONTACTS AND LOCATIONS:
Locations (1):
- Beni suef hospital, Banī Suwayf, Egypt